CLINICAL TRIAL: NCT04642599
Title: Bimanual Motor Skill Learning Through Robotics in Chronic Cerebellar Stroke Survivors and Healthy Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); Université Catholique de Louvain (Other); Louvain Bionics, UCLouvain (Unknown)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BimMSkL-Cerebellum
Record Dates: First submitted 2020-11-02; First posted 2020-11-24 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Cerebellar Stroke; Healthy Individuals (Controls)
Keywords: Stroke; Cerebellar Disorders; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Cerebellar Stroke; Cerebellar Hemorrhage; Cerebellar Infarction
MeSH Terms: conditions — Stroke; Cerebellar Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Evaluation of bimanual motor skill learning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic Cerebellar Stroke (Experimental): Participants with a chronic cerebellar stroke
  Interventions: Device: Bimanual motor skill learning with the REAplan® rehabilitation robot
- Healthy Individuals (Controls) (Active Comparator): healthy participants
  Interventions: Device: Bimanual motor skill learning with the REAplan® rehabilitation robot

INTERVENTIONS:
Device: Bimanual motor skill learning with the REAplan® rehabilitation robot — REAplan® rehabilitation robot: training to perform complex, coordinated, bimanual movements

SUMMARY:
To test capacity of chronic cerebellar stroke patients and healthy individuals to learn and retain a complex bimanual motor skill, trained on the neurorehabilitation robot REAplan® (bimanual version).

DETAILED DESCRIPTION:
Over 3 consecutive days, healthy individuals and chronic cerebellar stroke patients (1) will be evaluated and (2) will train on the neurorehabilitation robot REAplan®.

They will practice several tasks on the robot REAplan® (bimanual version), requiring either movements with the affected arm (unimanual tasks) or complex, coordinated movements with both arms (bimanual tasks).

In addition, several "classical" clinical scales and tests will be used to evaluate overall motor-sensory-cognitive functions (clinical tests, questionnaires, ...).

Hand/digits motor function will be also evaluated with the kinetic device DexTrain®.

ELIGIBILITY:
STROKE PATIENTS:

Inclusion Criteria:

* having a chronic cerebellar stroke (>6 months)
* aged 18-90 years
* with a demonstrated stroke (ischemic or hemorrhagic) lesion on brain imaging

Exclusion Criteria:

* difficulty in understanding or executing commands
* drug/alcohol abuse
* severe aphasia / cognitive deficits interfering with study
* inability to voluntarily move the affected arm (i.e. complete paralysis of the arm)
* multiple strokes / dementia / psychiatric condition

HEALTHY INDIVIDUALS:

Inclusion Criteria:

* 18-90 years

Exclusion Criteria:

* neurological conditions interfering with the study
* drug/alcohol abuse
* pyschiatric condition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in bi-SAT | Change between day 1 to 3
  Bimanual Speed/Accuracy Trade-off measured by the REAplan robot bimanual Speed/Accuracy Trade-off: mathematical computation of the relationship bewteen speed and accuracy
Change in bi-CO | Change between day 1 to 3
  Bimanual Coordination factor measured by the REAplan robot bimanual Coordination factor : mathematical measure of the phase coherence between velocities of both arms

SECONDARY OUTCOMES:
bi-SAT | Day 1 + day 3
  On bimanual REACHING (REAplan robot) bimanual Speed/Accurady Trade-off: mathematical computation of the relationship
bi-CO | Day 1 + day 3
  On bimanual REACHING (REAplan robot) bimanual Coordination factor: mathematical measure of the phase coherence between velocities of both arms
change in bi-Force | Change between day 1 to 3
  Bimanual forces : forces exerted in the wrong direction by each arm (Newtons)
bi-Force | Day 1 + day 3
  On bimanual REACHING (REAplan robot)
  bimanual forces : forces exerted in the wrong direction by each arm (Newtons)
bi-smoothness | Day 1+ day 3
  On bimanual REACHING (REAplan robot) Smoothness of movement : Spectral Arc Length (SPARC)
bi-error | Day 1 + day 3
  on bimanual REACHING (REAplan robot) Error in centimeters or degrees during bimanual reaching
Dextrain | Day 1 + day 3
  Kinetic device measuring the movements of each finger: error and co-activation (percentage)
Dextrain | Day 1 + day 3
  Kinetic device measuring the movements of each finger: speed (milliseconds)
Dextrain | Day 1 + day 3
  Kinetic device measuring the movements of each finger: force (Newton)
BBT | Day 1 + day 3
  Box & Blocks Test (timed transfert of blocks from one space to the other)
Modified International Cooperative Ataxia Rating Scale (MICARS) | Day 1
  Ataxia scale A high score describes strong ataxia and a low score describes weak ataxia
Fugl Meyer Upper extremity test | Day 2
  Tests impairments of the upper limb after stroke
Corsi block | Day 2
  Tests the visuo-spatial memory
Montreal Cognitive Assessment (MoCA) | Day 2
  Tests the short-term memory, visuospatial skills, executive functions, attention, concentration, working memory, language and orientation in time and space
Abilhand and activlim | Day 3
  Questionnaire about the bimanual hability during activities of the daily life

CONTACTS AND LOCATIONS:
Overall Officials: Yves Vandermeeren, MD, PhD, Principal Investigator — University Hospital of Mont-Godinne
Locations (1):
- CHU UCL Namur, Mont-Godinne, Neurology Department, Stroke Unit, Yvoir, Namur, Belgium

IPD SHARING:
Plan to Share IPD: Yes
the precise IPD plan has to be worked out in order to find the best public repository
Supporting Information: Study Protocol
Time Frame: Up to 2 years after publication of the scientific articles
Access Criteria: none (public)

REFERENCES:
- [Background] Yeganeh Doost M, Orban de Xivry JJ, Bihin B, Vandermeeren Y. Two Processes in Early Bimanual Motor Skill Learning. Front Hum Neurosci. 2017 Dec 20;11:618. doi: 10.3389/fnhum.2017.00618. eCollection 2017. PMID 29326573
- [Background] Dehem S, Gilliaux M, Lejeune T, Delaunois E, Mbonda P, Vandermeeren Y, Detrembleur C, Stoquart G. Effectiveness of a single session of dual-transcranial direct current stimulation in combination with upper limb robotic-assisted rehabilitation in chronic stroke patients: a randomized, double-blind, cross-over study. Int J Rehabil Res. 2018 Jun;41(2):138-145. doi: 10.1097/MRR.0000000000000274. PMID 29420360
- [Background] Doost MY, Orban de Xivry JJ, Herman B, Vanthournhout L, Riga A, Bihin B, Jamart J, Laloux P, Raymackers JM, Vandermeeren Y. Learning a Bimanual Cooperative Skill in Chronic Stroke Under Noninvasive Brain Stimulation: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2019 Jun;33(6):486-498. doi: 10.1177/1545968319847963. Epub 2019 May 15. PMID 31088342
- [Derived] Gathy E, Cadiat N, Gerardin E, Lambert J, Herman B, Leeuwerck M, Bihin B, Vandermeeren Y. Bimanual coordinated motor skill learning in patients with a chronic cerebellar stroke. Exp Brain Res. 2024 Jun;242(6):1517-1531. doi: 10.1007/s00221-024-06830-x. Epub 2024 May 9. PMID 38722346